| Pennsylvania State University, College of Medicine, | |
|---|---|
| Departme | Department of Family and Community Medicine Research |
| | Division |
| Official | HPV self-sampling among women at the PSH |
| Study Title | Colposcopy Clinics |
| Official | HRP-591 Protocol for Human Subject Research |
| Document | |
| Title | |
| Document | April 20, 2023 |
| date | |
| NCT | 04585243 |



# HRP-591 - Protocol for Human Subject Research

#### **Protocol Title:**

HPV self-sampling among women at the PSH colposcopy clinics

# **Principal Investigator:**

Name: Jennifer Moss, PhD

Department: Family & Community Medicine

Telephone: 717-531-0003 x 323429

E-mail Address: jmoss1@pennstatehealth.psu.edu

# **Version Date:**

April 22, 2021

#### Clinicaltrials.gov Registration #:

NCT04585243

#### **Important Instructions for Using This Protocol Template:**

This template is provided to help investigators prepare a protocol that includes the necessary information needed by the IRB to determine whether a study meets all applicable criteria for approval.

#### 1. **GENERAL INSTRUCTIONS:**

- Prior to completing this protocol, ensure that you are using the most recent version by verifying the
  protocol template version date in the footer of this document with the current version provided in the
  CATS IRB Library.
- Do not change the protocol template version date located in the footer of this document.
- Some of the items may not be applicable to all types of research. If an item is not applicable, please indicate as such or skip question(s) if indicated in any of the instructional text.

# • GRAY INSTRUCTIONAL BOXES:

- Type your protocol responses <u>below</u> the gray instructional boxes of guidance language. If the section or item is not applicable, indicate not applicable.
- Penn State College of Medicine/Penn State Health researchers: Delete the instructional boxes from the final version of the protocol prior to upload to CATS IRB (<a href="http://irb.psu.edu">http://irb.psu.edu</a>).
- Penn State researchers at all other campuses: Do NOT delete the instructional boxes from the final version of the protocol.
- Add the completed protocol template to your study in CATS IRB (<a href="http://irb.psu.edu">http://irb.psu.edu</a>) on the "Basic Information" page.

#### 2. CATS IRB LIBRARY:

Documents referenced in this protocol template (e.g. SOP's, Worksheets, Checklists, and Templates) can be
accessed by clicking the Library link in CATS IRB (<a href="http://irb.psu.edu">http://irb.psu.edu</a>).

### 3. PROTOCOL REVISIONS:

- When making revisions to this protocol as requested by the IRB, please follow the instructions outlined in the Study Submission Guide available in the Help Center in CATS IRB (<a href="http://irb.psu.edu">http://irb.psu.edu</a>) for using track changes.
- Update the Version Date on page 1 each time revisions are made.

If you need help...

**University Park and other campuses:** 

Office for Research Protections Human Research Protection Program

The 330 Building, Suite 205 University Park, PA 16802-7014

Phone: 814-865-1775 Fax: 814-863-8699 Email: <u>irb-orp@psu.edu</u> **College of Medicine and Penn State Health:** 

**Human Subjects Protection Office** 

90 Hope Drive, Mail Code A115, P.O. Box 855

Hershey, PA 17033

(Physical Office Location: Academic Support Building

Room 1140)

Phone: 717-531-5687 Email: <u>irb-hspo@psu.edu</u>

#### **Table of Contents**

21.0

22.0

References

**Confidentiality, Privacy and Data Management** 

| 1.0 | Objectives |
|---|---|
| 2.0 | Background |
| 3.0 | Inclusion and Exclusion Criteria |
| 4.0 | Recruitment Methods |
| 5.0 | Consent Process and Documentation |
| 6.0 | HIPAA Research Authorization and/or Waiver or Alteration of Authorization |
| 7.0 | Study Design and Procedures |
| 8.0 | Subject Numbers and Statistical Plan |
| 9.0 | Data and Safety Monitoring Plan |
| 10.0 | Risks |
| 11.0 | Potential Benefits to Subjects and Others |
| 12.0 | Sharing Results with Subjects |
| 13.0 | Subject Payment and/or Travel Reimbursements |
| 14.0 | Economic Burden to Subjects |
| 15.0 | Resources Available |
| 16.0 | Other Approvals |
| 17.0 | Multi-Site Study |
| 18.0 | Adverse Event Reporting |
| 19.0 | Study Monitoring, Auditing and Inspecting |
| 20.0 | Future Undetermined Research: Data and Specimen Banking |

# 1.0 Objectives

# 1.1 Study Objectives

The main objective is to compare the test characteristics of the human papillomavirus (HPV) self-sampling kit versus clinician-sampled HPV testing for cervical cancer screening. This study seeks to find out if the HPV self-sampling kit is non-inferior to standard clinician-sampling practices.

# 1.2 Primary Study Endpoints

The primary outcomes of this study are to analyze the screening results on self-sampling kits compared to clinician-collected HPV test, Pap smear results, and colposcopy.

# 1.3 Secondary Study Endpoints

Secondary endpoints will include acceptability of self-sampling and barriers to cervical cancer screening. These endpoints will be analyzed to try to circumvent barriers to the cervical cancer screening and ascertain whether self-sampling is a viable alternative.

# 2.0 Background

#### 2.1 Scientific Background and Gaps

The American Cancer Society estimates that 4,170 women in the United States (US) will die from cervical cancer in 2018. Screening can reduce cancer mortality by (1) detecting malignancies when they are more treatable and (2) for some tests, identifying precancerous lesions for removal. Guidelines recommend cytology and/or HPV testing for cervical cancer screening among women ages 30-65 years, but screening rates are suboptimal. 3, 4

To help bridge these gaps in screening, HPV self-sampling would be an alternative to clinical screening. However, there are concerns about the efficacy and comparability of self-sampling kits as an effective tool to detect cervical cancer.

#### 2.2 Previous Data

There have been previous studies about the effectiveness of self-collected samples as an alternative to clinician collected samples. Some studies state that HPV testing is more sensitive than Pap testing.<sup>5</sup> There is a possibility that these to samples have similar sensitivity.<sup>6</sup> Based on this information, examining test characteristics and acceptability of each technique is necessary to support larger efforts to make self-sampling available.

# 2.3 Study Rationale

The impact of the proposed project is to compare HPV self-screening results with Pap smear results, clinician-collected HPV test, and colposcopy to ultimately improve the uptake of HPV screening.

# 3.0 Inclusion and Exclusion Criteria

#### 3.1 Inclusion Criteria

- 1. Ages 30-65 years
- 2. Penn State Health (PSH) patient
- 3. Female
- 4. Has an intact cervix
- 5. With abnormal findings on Pap/HPV test that requires a colposcopy for follow-up
- 6. Speaks, reads, or writes well in English or Spanish

#### 3.2 Exclusion Criteria

- 1. Pregnant
- 2. Cognitively impaired
- 3. Incarcerated
- 4. Complete hysterectomy
- 5. History of cervical treatment for abnormal Pap/HPV test (i.e., cryotherapy, Loop electrosurgical excision procedure(LEEP))

# 3.3 Early Withdrawal of Subjects

# 3.3. 1 Criteria for removal from study

If the subjects becomes pregnant or does not complete the study activities they will be removed from the study.

### 3.3. 2 Follow-up for withdrawn subjects

The withdrawal will be documented and the subject will be replaced if the timeline allows.

#### 4.0 Recruitment Methods

# 4.1 Identification of subjects

Potential participants will be identified from participating Family and Community Medicine (FCM) and OBGYN clinics at Penn State Health when they are determined to have abnormal findings on Pap/HPV test that requires a colposcopy for follow-up. Potential participants will be identified in one of three ways:

- (1) A member of the study team will access the electronic medical records (EMR) for Dr. Ramirez's and Dr. Wright's OBGYN patients that meet the study criteria and have an upcoming colposcopy appointment. Then, a member of the study team will call the participant about possible involvement in the study.
- (2) Clinicians will provide general information (via recruitment cards) about the study during the colposcopy appointment (if the patient was not previously contacted or was scheduled less than two weeks from their appointment). Patients will be advised to contact the study team using the information on the card if interested in participating.
- (3) After a patient's appointment, if the clinician believes the individual could meet eligibility criteria for the study, the clinician will send the contact information for these patients to the study team members

through a secure message in the Electronic Medical Record. For this option, patients would not have been presented with the research opportunity during their appointment; clinicians may not have had a recruitment card available to give to their patient or may simply have forgotten to share the study opportunity.

# 4.2 Recruitment process

# 4.2. 1 How potential subjects will be recruited.

Clinicians will identify potential participants they think would be eligible for the study and provide some general information (via the recruitment cards) to the participants. Members of the study team (non-clinical staff) will prospectively review clinic schedules in order to identify potential participants, and clinicians may also identify patients after their scheduled appointment. This will ensure that enrollment numbers are met and that all potentially eligible participants are provided with a recruitment card by their clinician or contacted directly by a study team member.

# 4.2. 2 Where potential subjects will be recruited.

Potential subject will be recruited from Penn State Health Family & Community Medicine and OBGYN clinics.

# 4.2. 3 When potential subjects will be recruited.

Participants will be recruited at their colposcopy appointment in the clinician's office or over the phone by a study team member. The participant will be screened for eligibility and provide verbal implied consent.

4.2. 4 Describe the eligibility screening process and indicate whether the screening process will occur before or after obtaining informed consent. Screening begins when the investigator obtains information about or from a prospective participant in order to determine their eligibility. In some studies, these procedures may not take place unless HIPAA Authorization is obtained OR a waiver of HIPAA Authorization when applicable for the screening procedures is approved by the IRB. [For FDA regulated studies, consent for any screening activities would need to be obtained prior to screening unless specifically waived by the IRB.]

Initial screening may occur before obtaining implied consent. A member of the research team will review the EMR for FCM/ OBGYN patients that meet the study criteria. Then a study team member will call the person to complete the screening process and then obtain verbal consent. A study team member will mail the participant the study materials and a summary explanation of research.

# 5.0 Consent Process and Documentation

| 5.1 | Consent Process: |
|---|---|
| | Check all applicable boxes below: |
| | Informed consent will be sought and documented with a written consent form [Complete Sections |
| | 5.2 and 5.6] |

| | Informed consent will be sought but some of the elements of informed consent will be omitted or altered (e.g., deception). [Complete section 5.2, 5.4 and 5.6] |
|---|---|
| | ☐ Informed consent will not be obtained – request to completely waive the informed consent requirement. [Complete Section 5.5] |
| Γhe f | ollowing checkbox is for all locations EXCEPT Penn State Health and College of Medicine: |
| | Exempt Research at all Locations Except Penn State Health and the College of Medicine: If you believe that the research activities outlined meet one or more of the criteria outlined in "HRP-312-Worksheet- Exemption Determination." Please verify by checking this box that if conducting an exempt research study, the consent process will disclose the following (all of which are included in "HRP-590- Consent Guidance for Exempt Research"): Penn State affiliation; name and contact information for the researcher and advisor (if the researcher is a student); the activities involve research; the procedures to be performed; participation is voluntary; that there are adequate provisions to maintain the privacy interests of subjects and the confidentiality of the data; and subjects may choose not to answer specific |
| | questions. |

Note: If this box has been checked, skip the remainder of section 5 and proceed to section 6 of this protocol. If the investigator's assessment is inaccurate, an IRB Analyst will request revision to the protocol and that an informed consent form be submitted for review and approval. Except for exemptions where Limited IRB Review (see "HRP-312- Worksheet- Exemption Determination") is

required or where otherwise requested by the IRB, informed consent forms for research activities

determined to be exempt without Limited IRB Review are generally not required to be submitted for review and approval by the University Park IRB.

#### **5.2** Obtaining Informed Consent

#### 5.2. 1 Timing and Location of Consent

Participants will be consented up to 21 days before or after their colposcopy appointment over the phone and answers will be input into REDCap by a member of the study team. Once the participant has been screened and gives verbal consent, participants will be mailed a paper copy of the summary explanation of research with the HPV self-sampling kit.

# 5.2. 2 Coercion or Undue Influence during Consent

After a review of the research study via the Summary Explanation of Research, subjects will be asked if they give consent to participate in the survey. Subjects will be reminded that they may refuse to answer any question and end their participation at any time, and their decision on whether or not to participate in this research will not affect their medical care.

#### 5.3 Waiver of Written Documentation of Consent

| | | | The research presents no more that minimal risk of harm to subjects and involves no procedures for which written consent is normally required outside of the research context. |
|---|---|---|---|
| | | | The only record linking the subject and the research would be the consent document and the principal risk would be potential harm resulting from a breach of confidentiality. Each subject will be asked whether the subject wants documentation linking the subject with the research, and the subject's wishes will govern. (Note: This condition is not applicable for FDA-regulated research. If this category is chosen, include copies of a consent form and /or parental permission form for participants who want written documentation linking them to the research.) |
| | | | If the subjects or legally authorized representatives are members of a distinct cultural group or community in which signing forms is not the norm, that the research presents no more than minimal risk of harm to subjects and provided there is an appropriate alternative mechanism for documenting that informed consent was obtained. ( <i>Note: This condition is not applicable for FDA-regulated research.</i> ) |
| | | | Describe the alternative mechanism for documenting that informed consent was obtained: |
| | 5.3. | 2 | Indicate what materials, if any, will be used to inform potential subjects about the research (e.g., a letter accompanying a questionnaire, verbal script, implied consent form, or summary explanation of the research) |
| | | | Verbal script (including summary explanation of the research) |
| 5.4 | | | ed consent will be sought but some of the elements of informed consent will be omitted or (e.g., deception). |
| | 5.4. | 1 | Indicate the elements of informed consent to be omitted or altered |
| | | | Not applicable. |
| | 5.4. | 2 | Indicate why the research could not practicably be carried out without the omission or alteration of consent elements |
| | | | Not applicable. |
| | 5.4. | 3 | Describe why the research involves no more than minimal risk to subjects. |
| | | | Not applicable. |
| | 5.4. | 4 | Describe why the alteration/omission will not adversely affect the rights and welfare of subjects. |

**5.3.** 1 Indicate which of the following conditions applies to this research:

Not applicable.

5.5

5.6

| 5.4. 5 | If the research involves using identifiable private information or identifiable biospecimens, describe why the research could not be practicably be carried out without using such information or biospecimens in an identifiable format. |
|---|---|
| | Not applicable. |
| 5.4. 6 | Debriefing |
| | Not applicable. |
| Inform<br>require | ed consent will not be obtained – request to completely waive the informed consent ement |
| 5.5. 1 | Indicate why the research could not practicably be carried out without the waiver of consent |
| | Not applicable. |
| 5.5. 2 | Describe why the research involves no more than minimal risk to subjects. |
| | Not applicable. |
| 5.5. 3 | Describe why the alteration/omission will not adversely affect the rights and welfare of subjects. |
| | Not applicable. |
| 5.5. 4 | If the research involves using identifiable private information or identifiable biospecimens, describe why the research could not be practicably be carried out without using such information or biospecimens in an identifiable format. |
| | Not applicable. |
| 5.5. 5 | Additional pertinent information after participation |
| | Not applicable. |
| Conser | nt – Other Considerations |

# 5.6. 1 Non-English-Speaking Subjects

The study will include Spanish-speaking participants. Staff who speak Spanish fluently will communicate with these subjects during the study procedures. Alternatively, if the preferred language is Spanish, LanguageLine can be utilized for translation.

| 5. | 6. | 2 | Cognitively | / Impaired Adults |
|----|----|---|-------------|-------------------|

**5.6.2.1** Capability of Providing Consent

Not applicable.

5.6.2.2 Adults Unable to Consent

Not applicable.

5.6.2.3 Assent of Adults Unable to Consent

Not applicable.

- 5.6. 3 Subjects who are not yet adults (infants, children, teenagers)
  - 5.6.3.1 Parental Permission

Not applicable.

5.6.3.2 Assent of subjects who are not yet adults

Not applicable.

- 6.0 HIPAA Research Authorization and/or Waiver or Alteration of Authorization
  - 6.1 Authorization and/or Waiver or Alteration of Authorization for the Uses and Disclosures of PHI

| Check a | All that apply: Not applicable, no identifiable protected health information (PHI) is accessed, used or disclosed in this study. [Mark all parts of sections 6.2 and 6.3 as not applicable] |
|---|---|
| | Authorization will be obtained and documented as part of the consent process. [If this is the only box checked, mark sections 6.2 and 6.3 as not applicable] |
| $\boxtimes$ | Partial waiver is requested for recruitment purposes only (Check this box if patients' medical records will be accessed to determine eligibility before consent/authorization has been obtained). [Complete all parts of sections 6.2 and 6.3] |
| | Full waiver is requested for entire research study (e.g., medical record review studies). [Complete all parts of sections 6.2 and 6.3] |
| $\boxtimes$ | Alteration is requested to waive requirement for written documentation of authorization (verbal authorization will be obtained). [Complete all parts of sections 6.2 and 6.3] |

#### 6.2 Waiver or Alteration of Authorization for the Uses and Disclosures of PHI

# 6.2. 1 Access, use or disclosure of PHI representing no more than a minimal risk to the privacy of the individual

# 6.2 .1.1 Plan to protect PHI from improper use or disclosure

Information is included in the "Confidentiality, Privacy, and Data Management" section of this protocol.

# 6.2 .1.2 Plan to destroy identifiers or a justification for retaining identifiers

Protected health information (PHI) will be used for recruitment through the EMR by members of the study team. All EMR data and study data will be input into REDCap (i.e., insurance status, and date and results of previous Pap/HPV tests). There will be two databases for participant data. The first linking list will contain the medical record number (MRN) and the unique study ID number. This list will be destroyed after data collection. The second linking list will have the study ID with all study data. This second linking list will be kept for up to two years after data collection.

Identifiers will be destroyed after the completion of data analysis.

# 6.2. 2 Explanation for why the research could not practicably be conducted without access to and use of PHI

The proposed study requires enrollment of participants who have abnormal findings on Pap/HPV tests to compare those results with the findings from a self-sampled HPV test. Identification of these participants would be infeasible using other methods.

# 6.2. 3 Explanation for why the research could not practicably be conducted without the waiver or alteration of authorization

Prospective identification of participants with abnormal findings on Pap/HPV tests using PHI prior to consent will be more practical and efficient than obtaining consent prior to determining whether a potential participant had abnormal findings on these tests.

Having participants provide implied consent by using the Summary Explanation of Research Is more practical because it allows the study team to send a kit to participants prior to their appointment, and therefore gives the participant more time to complete study procedures. This process also makes it easier to participate in the study since all materials are mailed to the participants home, and they will not take up any extra clinic time during their appointment.

#### 6.3 Waiver or alteration of authorization statements of agreement

Protected health information obtained as part of this research will not be reused or disclosed to any other person or entity, except as required by law, for authorized oversight of the research study, or for other permitted uses and disclosures according to federal regulations.

The research team will collect only information essential to the study and in accord with the 'Minimum Necessary' standard (information reasonably necessary to accomplish the objectives of the research) per federal regulations.

Access to the information will be limited, to the greatest extent possible, within the research team. All disclosures or releases of identifiable information granted under this waiver will be accounted for and documented.

# 7.0 Study Design and Procedures

# 7.1 Study Design

After the participant is screened and informs the study team member that they would like to enroll in the study, an HPV self-sampling kit, the instructions on how to use it, a summary explanation of research, PSH lab Pathology Services Special Account Requisition form, and a letter from the principal investigator (PI) (see "Moss Self-sampling Letter") will be mailed to study participants. Participants will be asked to complete the HPV self-sampling kit within a week. 3-5 days before the colposcopy appointment a study team member will reach out to check if study participants have completed their HPV self-sampling kit. Those that have completed the kit will complete a survey (HPVSelfSamplingAcceptabilityAn) over the phone and get an appointment reminder. They will mail their HPV self-sampling kit and PSH lab Pathology Services Special Account Requisition form to the lab. On the day of their appointment, their clinician will perform a colposcopy following normal clinical procedures.

Participants who have not completed their HPV self-sampling kit will get instructions not to use the HPV self-sampling kit before the colposcopy and get an appointment reminder. They will then go to their appointment where the clinician will perform the colposcopy. After their visit, the participant will receive a reminder to use the HPV self-sampling kit within two weeks. The participant will receive a maximum of three phone calls after their colposcopy appointment to remind them to return their completed self-sampling kit. Seven days after the colposcopy appointment the research project manager will call the participant to determine if she completed the HPV self-sampling kit and, if so, they will complete a survey (HPVSelfSamplingAcceptabilityAn) over the phone. If the participant has not completed the kit or does not respond, a second phone call will then occur 10 days after the colposcopy appointment. A final phone call will up to 21 days after the colposcopy appointment. If the self-sampling kit is not collected 21 days after the colposcopy or if the study team is unable to reach the participant, their participation will be considered incomplete.

Participants must complete the self-sampling kit within 14 days before or after their colposcopy visit, meaning that there is a 28 day window for participants to collect the sample. A 2<sup>nd</sup> HPV self-sampling kit will only be mailed if the participant states that she lost or did not receive the first one. Participants will receive a maximum of 2 HPV self-sampling kits.

Once the HPV self-sampling kit has been returned and the survey completed, the study participants will be mailed an incentive in the form of a Greenphire ClinCard, and a thank you letter from the PI. Analysis of the self-sampling specimens will be conducted to determine HPV DNA positivity to compare to the results of the previous Pap test, HPV test, and colposcopy. EMR data will be used to check insurance status, and the date and result of Pap test, HPV test, and colposcopy.

# 7.2 Study Procedures

Survey and HPV self-sampling kit

# 7.2. 1 Up to 21 days before the colposcopy appointment

A study team member will obtain implied verbal consent from the participants and mail the HPV self-sampling kit with the instructions, a summary explanation of research, PSH lab Pathology Services Special Account Requisition form, and Moss Self-sampling Letter.

# 7.2. 2 3-5 days before the colposcopy appointment

A study team member will call study participants to provide a reminder to attend their colposcopy appointment and, if they completed their HPV self-sampling kit, take a survey (HPVSelfSamplingAcceptabilityAn) over the phone. Those that did not complete the HPV self-sampling kit will get an appointment reminder and be told not to use the self-sampling kit before the colposcopy.

# 7.2. 3 Up to 21 days after colposcopy appointment

Seven days after their colposcopy visit, a study team member will call those participants who did not complete the HPV self-sampling kit prior to the colposcopy appointment to complete a survey (HPVSelfSamplingAcceptabilityAn) over the phone. If they still have not completed the HPV self-sampling kit, they will be reminded to complete the self-sampling kit and a study team member will schedule another phone call to complete the survey (HPVSelfSamplingAcceptabilityAn) up to 21 days post-colposcopy. Once the HPV self-sampling kit has been returned and the survey completed, the study team will mail out the participant's incentive and the Thank You Letter. If the participant did not complete the kit then no further contact will be made after day 21, and the participant will not receive a gift card nor will they be included in the goal of 30 total completers.

# 7.3 Duration of Participation

Participants will be in the study for up to five weeks.

# 7.4 Test Article(s) (Study Drug(s) and/or Study Device(s))

# 7.4. 1 Description

The Evalyn® Brush is a self-sampling kit that screens for HPV, a leading cause of cancer death among women. This tool has recently been FDA approved, but has not been incorporated into national clinical guidelines. This product is a small pink capped brush that can be used to take a sample of cervical cells.

#### 7.4. 2 Treatment Regimen

Participants will take a sample of their cervix cells that amounts to a few millimeters of bio specimen.

# 7.4. 3 Method for Assigning Subject to Treatment Groups

Not applicable

#### 7.4. 4 Subject Compliance Monitoring

Subject compliance will be confirmed once their lab results are received from the PSH lab.

# 7.4. 5 Blinding of the Test Article

Not applicable

# 7.4. 6 Receiving, Storage, Dispensing and Return

# 7.4 .6.1 Receipt of Test Article

1 HPV self-sampling kit will be sent to the PSH lab in a prepaid mailing. Inside the mailing will be the HPV self-sampling kit with the instructions and a PSH lab Pathology Services Special Account Requisition form. The kits will be supplied by the Department of Family and Community Medicine.

# 7.4 .6.2 Storage

Before HPV self-sampling kits are sent to study participants, they will be stored in a locked cabinet in the Department of Family and Community Medicine offices at 134 Sipe Ave. Kits mailed to the lab will be disposed of after analysis.

# 7.4 .6.3 Preparation and Dispensing

Before it is sent to the participant, the PSH lab Pathology Services Special Account Requisition document will be labeled with the participant's ID #, date of birth, and sex. The Mailing will include the HPV self-sampling kit with the instructions, a summary explanation of research, PSH lab Pathology Services Special Account Requisition form and Moss\_Self-sampling Letter. Also, the package will include a prepaid and labeled mailing to send the kit and Pathology Services Special Account Requisition document to the PSH lab. Participants will need to include the date and time of sample collection on the Requisition form.

# 7.4 .6.4 Return or Destruction of the Test Article

HPV self-sampling kits not be returned to participants. The samples will be analyzed and the kits will be destroyed by the PSH lab once analysis is complete.

### 7.4 .6.5 Prior and Concomitant Therapy

Not applicable

# 8.0 Subject Numbers and Statistical Plan

# 8.1 Number of Subjects

We expect to consent and screen no more than 60 women to achieve a final sample size of 30 participants after accounting for potential screen failures.

# 8.2 Sample size determination

Assuming p<.05 and beta>0.80, we need 30 participants to determine concordance/non-inferiority of test results across the two different methods using a Fisher's exact test and Cohen's kappa coefficient.

#### 8.3 Statistical methods

We will conduct Fisher's exact tests to examine our primary study outcome, i.e., concordance/noninferiority of HPV self-sampling test results versus clinician-sampled test results. Additional analyses of the concordance across test will use Cohen's kappa coefficient. In addition, we will summarize survey results using descriptive analysis, including calculating means, Pearson's correlation coefficients, and Fisher's exact tests.

| | | Tible 3 chact tests. |
|-----|---------|--------------------------------------------|
| 9.0 | Data aı | Data and Safety Monitoring Plan |
| | 9.1 | Periodic evaluation of data |
| | | Not applicable. |
| | 9.2 | Data that are reviewed |
| | | Not applicable. |
| | 9.3 | Method of collection of safety information |
| | | Not applicable. |
| | 9.4 | Frequency of data collection |
| | | Not applicable. |
| | 9.5 | Individuals reviewing the data |
| | | Not applicable. |
| | 9.6 | Frequency of review of cumulative data |
| | | Not applicable. |
| | 9.7 | Statistical tests |
| | | Not applicable. |

#### 9.8 Suspension of research

Not applicable.

#### **10.0** Risks

Potential risks associated with this research are minimal. Loss of confidentiality is a risk of participation. All information entered into REDCap will be password protected with limited access to specific members of the study team. There may also be risks from participants misusing the self-sampling kit. This may cause minor discomfort if used improperly.

# 11.0 Potential Benefits to Subjects and Others

# 11.1 Potential Benefits to Subjects

None

#### 11.2 Potential Benefits to Others

Understanding how the results of the HPV self-sampling kit compare to clinician-collected HPV tests, Pap smears, and colposcopies will ultimately help to create a better screening process. If the findings are similar across tests, HPV self-sampling may emerge as an effective option for cervical cancer screening among underserved populations without routine access to preventive healthcare.

# **12.0** Sharing Results with Subjects

Not applicable.

# **13.0** Subject Payment and/or Travel Reimbursements

\$15 via Greenphire ClinCard. After the participant completes the follow-up survey they will be asked to provide the information necessary in order to set up the Greenphire Clincard. Once the study team receives confirmation that their completed kit was received by PSH, the study team will mail the clincard to the participant at their preferred address along with the thank you letter.

# 14.0 Economic Burden to Subjects

#### 14.1 Costs

Not applicable

#### 14.2 Compensation for research-related injury

Not applicable

#### **15.0** Resources Available

#### 15.1 Facilities and locations

Participants will be identified from participating Family and Community Medicine and OBGYN clinics at PSH when they are determined to have abnormal findings on Pap/HPV test that requires a colposcopy for follow-up. Physicians will perform the colposcopy per standard clinical guidelines. Self-sampling kits will be mailed into a PSH lab for analysis with supplies given by the study team. Afterwards, a study team member will collect survey data from participants over the phone.

# 15.2 Feasibility of recruiting the required number of subjects

Among the PSH study clinics, at least 18 potentially-eligible patients receive a colposcopy each month. All potentially-eligible patients will be invited to join the study, and they will be screened and consented if there are eligible. 30 subjects will be enrolled into the study. Among the 120 invited to participate in this study, we expect 50% (60) to agree to participate and meet eligibility. This should provide a large enough sample size to obtain 30 participants who complete all study procedures. Based on these figures, it will take approximately 7 months to invite 120 subjects and enroll 30 participants who complete all study procedures.

# 15.3 PI Time devoted to conducting the research

The PI will use dedicated research time to conduct this research.

#### 15.4 Availability of medical or psychological resources

Not applicable.

#### 15.5 Process for informing Study Team

The research team will meet regularly to discuss this study, its procedures, and any issues that may arise.

# **16.0** Other Approvals

# 16.1 Other Approvals from External Entities

Not applicable.

# 16.2 Internal PSU Committee Approvals

| Che | eck all that apply: |
|---|---|
| | Anatomic Pathology – <b>Penn State</b> Health <b>only</b> – Research involves the collection of tissues or use of pathologic specimens. Upload a copy of "HRP-902 - Human Tissue For Research Form" in CATS IRB. |
| | Animal Care and Use – <b>All campuses</b> – Human research involves animals and humans or the use of human tissues in animals |

| | | in a PSU research lab, biological toxins, carcinogens, infectious agents, recombinant viruses or DNA or gene therapy). |
|---|---|---|
| | | Clinical Laboratories – <b>Penn State Health only</b> – Collection, processing and/or storage of extra tubes of body fluid specimens for research purposes by the Clinical Laboratories; and/or use of body fluids that had been collected for clinical purposes but are no longer needed for clinical use. Upload a copy of "HRP-901 - Human Body Fluids for Research Form" in CATS IRB. |
| | | Clinical Research Center (CRC) Advisory Committee – <b>All campuses</b> – Research involves the use of CRC services in any way. |
| | | Conflict of Interest Review – All campuses – Research has one or more of study team members indicated as having a financial interest. |
| | | Radiation Safety – <b>Penn State Health only</b> – Research involves research-related radiation procedures. All research involving radiation procedures (standard of care and/or research-related) must upload a copy of "HRP-903 - Radiation Review Form" in CATS IRB. |
| | | IND/IDE Audit – All campuses – Research in which the PSU researcher holds the IND or IDE or intends to hold the IND or IDE. |
| | | Scientific Review – <b>Penn State Health only</b> – All investigator-written research studies requiring review by the convened IRB must provide documentation of scientific review with the IRB submission. The scientific review requirement may be fulfilled by one of the following: (1) external peer-review process; (2) department/institute scientific review committee; or (3) scientific review by the Clinical Research Center Advisory committee. NOTE: Review by the Penn State Health Cancer Institute (PSCI) Protocol Review Committee or the PSCI Disease Team is required if the study involves cancer prevention studies or cancer patients, records and/or tissues. For more information about this requirement see the IRB website. |
| 17.0 | Multi- | Site Study |
| | 17.1 | Other sites |
| | | Not applicable. |
| | 17.2 | Communication Plans |
| | | Not applicable. |
| | 17.3 | Data Submission and Security Plan |
| | | Not applicable. |
| | 17.4 | Subject Enrollment |
| | | Not applicable. |

# 17.5 Reporting of Adverse Events and New Information

Not applicable.

# 17.6 Audit and Monitoring Plans

Not applicable.

# 18.0 Adverse Event Reporting

# 18.1 Reporting Adverse Reactions and Unanticipated Problems to the Responsible IRB

In accordance with applicable policies of The Pennsylvania State University Institutional Review Board (IRB), the investigator will report, to the IRB, any observed or reported harm (adverse event) experienced by a subject or other individual, which in the opinion of the investigator is determined to be (1) unexpected; and (2) probably related to the research procedures. Harms (adverse events) will be submitted to the IRB in accordance with the IRB policies and procedures.

# 19.0 Study Monitoring, Auditing and Inspecting

# 19.1 Auditing and Inspecting

The investigator will permit study-related monitoring, audits, and inspections by the Penn State quality assurance program office(s), IRB, the sponsor, and government regulatory bodies, of all study related documents (e.g., source documents, regulatory documents, data collection instruments, study data etc.). The investigator will ensure the capability for inspections of applicable study-related facilities (e.g., pharmacy, diagnostic laboratory, etc.).

# 20.0 Future Undetermined Research: Data and Specimen Banking

# 20.1 Data and/or specimens being stored

Not Applicable

# 20.2 Location of storage

Not Applicable

# 20.3 Duration of storage

Not Applicable

#### 20.4 Access to data and/or specimens

Not Applicable

# 20.5 Procedures to release data or specimens

Not Applicable

# 20.6 Process for returning results

Not Applicable

# 21.0 References

- 1. Siegel, RL, Miller, KD, Jemal, A. Cancer statistics, 2018. CA Cancer J Clin 2018;68(1):7-30.
- 2. Shieh, Y, Eklund, M, Sawaya, GF, et al. Population-based screening for cancer: hope and hype. Nature Reviews Clinical Oncology 2016.2.
- 3. U. S. Preventive Services Task Force. Final recommendation statement: Cervical cancer: Screening; 2018.
  - https://www.uspreventiveservicestaskforce.org/Page/Document/RecommendationStatementFinal/cervical-cancer-screening2. Accessed 2018.
- 4. Saslow, D, Solomon, D, Lawson, HW, et al. American Cancer Society, American Society for Colposcopy and Cervical Pathology, and American Society for Clinical Pathology screening guidelines for the prevention and early detection of cervical cancer. CA Cancer J Clin 2012;62(3):147-172.
- 5. Mayrand, Marie-Helene, Duarte-Franco, Aliane, Rodrigues, Isabel, Walter, Stephen, Hanley, James, Ferenczy, Alex, Ratman, Sam, Coutlee, Franciis, Franco, Eduardo. Human Papillomavirus DNA versus Papanicolaou Screening Tests for Cervical Cancer. The New England Journal of Medicine
- 6. Polman, Nicole, Ebisch, Renee, Heideman, Danielle, Melchers, Willem, Bekkers, Ruud, Molijn, Anco, et al. Performance of human papillomavirus testing on self-collected versus clinician-collected samples for the detection of cervical intraepithelial neoplasia of grade 2 or worse: a randomised, paired screen-positive, non-inferiority trial. The Lancet Oncology's 2019, 20(2): 229-238.